CLINICAL TRIAL: NCT01368679
Title: Phase III of the Prospective, Non-randomized and Multicenter Clinical Evaluation of the Safety and Performance of the Modular AAA Stent-Graft System When Used in the Treatment of Subjects With Abdominal Aortic Aneurysms (AAA)
Brief Title: A Clinical Study to Evaluate the Safety and Performance of the Modular AAA Stent-Graft System
Acronym: Stent-Graft
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Scitech Produtos Medicos Ltda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Scitech 003
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Cardiovascular Diseases; Abdominal Aortic Aneurysm
Keywords: Aortic Aneurysm, Abdominal; Abdominal Aortic
MeSH Terms: conditions — Cardiovascular Diseases; Aortic Aneurysm, Abdominal | interventions — Stents; Endovascular Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endoprothesis Scitech (Experimental): The endoprothesis of SCITECH is a self-expandable stent mixed (laser cut and wire plotted) covered with polyester fabric. The delivery system has lower profile than the existing market and this approach allows the passage of the delivery system through the femoral artery with ease and without dissection. Fixation has proximal and distal securing lower rates of leakage and displacement.
  The delivery system is done by linear drive or screw diameters greater than 30mm
  Interventions: Procedure: Endoprothesis Implantation

INTERVENTIONS:
Procedure: Endoprothesis Implantation — stent implantation in the abdominal artery using endovascular
  Other Names: stenting; endovascular procedure

SUMMARY:
This is a prospective multicenter observational study with 20 patients to evaluate the performance of SCITECH stent for treatment of AAA. Will be enrolled the patient demographics, laboratory tests, medical history, clinical evaluation, physical examination, adverse events.

The benefits and risks of the study should be explained before any specific test or procedure of the study. The written consent must be obtained from the patient. No action specifies the study should be performed while the patient has not signed the form of consent.

DETAILED DESCRIPTION:
Until the 90s the treatment of AAA was exclusively surgical, presenting a significant risk of death, however, many patients could not undergo this surgery because of the invasive nature of the procedure.

The mortality and comorbidity were associated with significant surgical repair of AAAs, particularly in elderly patients with multiple medical problems. Surgical complications were mainly associated with the surgical incision, comorbidity presented by the patient, changes cardiopulmonary and problems related to clotting of the patient. The postoperative complications included bleeding, renal failure, paraplegy, and the need for prolonged ventilatory support. The literature shows that mortality rates for elective surgery is 0-6.1%, with 2.7% as average.

Due to the risks and complexities inherent in surgical procedures, various devices and alternative methods have been proposed to treat aneurysms. The method most used today is the implantation of stents through a delivery system. This method is defined as minimally invasive to dispense the need for opening the abdominal cavity through large incisions, and use a remote access (common femoral artery or external iliac) to introduce and deploy the device via an endovascular route.

With technological progress have been developed many devices, all with similar characteristics, which are currently used in different countries. Numerous devices are currently used to treat aneurysms.

Over the past 10 years, were developed and approved new stents, however, despite the advances that have represented the use of minimally invasive devices, and evidence of improvement in indices of morbidity and mortality in the first six months, there is still a need to improve results, since the long-term endovascular treatment is equal to the conventional surgical treatment. With the technological devices you can improve your long-term performance and obviate the need for dissection of the femoral vessels using thinner delivery devices that allow percutaneous introduction.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years
2. Concordance of the patient through the end of a written consent form approved by the local Ethics Committee;
3. Proximal colon with the following characteristics: the intima to intima diameter of 16 to 30mm; Length of the proximal neck greater than 8mm angulation of the aorta justarenal less than or equal to 60 degrees.
4. Iliac axes: the distal neck length greater than 10mm; the intima to intima diameter between 7 and 20mm.
5. Present at least one of the following:

   * Aneurysm diameter > 4.5 cm,
   * Aneurysm that has increased in size from 0.5cm in the last six months,
   * aneurysm with maximum diameter greater at least one and half times the expected normal aortic diameter.
6. Patient who has access to the iliac or femoral artery for stent implantation in the abdominal aorta.
7. The patient is able to meet the follow-up examination in 30 days, 180 days and 360 days.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with dissecting aneurysm.
3. Patients with acute symptoms of ruptured aneurysm.
4. Patient with acute vascular injury.
5. Patients referred for emergency treatment.
6. Patients with tortuous iliac / femoral exceedingly difficult to access.
7. Patient with abdominal aortic dissection.
8. Patient with congenital anomalies after the placement of the stent will cause the main blood flow occlusion.
9. The patient with unstable angina.
10. Morbid obesity, or other clinical conditions that severely inhibit visualization of the USG of the aorta.
11. Patient with a history of connective tissue disease syndrome (eg, Marfan or Ehler's-Danlos syndrome).
12. Patient with a history of bleeding with the refusal of blood transfusions.
13. Patients with known hypersensitivity to the means of anticoagulation or contrast.
14. Patient with chronic renal failure (creatinine increase greater than or equal to 2.0 mg / dL).
15. Mycotic aneurysm or a systemic infection activates
16. Patient with a known allergy or intolerance to the components of these devices.
17. Patient is currently participating in another clinical trial investigating whether the device or drug.
18. Patient with other medical observations, social or psychological, according to the investigator's opinion, impossible to receive this treatment, the procedures and continuation of the pre and post-treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Evaluation of Adverse Events | Adverse Events
  * Evaluate the serious adverse events at 30 days after the implant the stent.
  * Evaluate safety of this stent for treatment of AAA after 30, 180 and 360 days implant.

SECONDARY OUTCOMES:
Evaluation the performance of the stent delivery system | Performance of stent-grift
  Evaluate the performance of the stent delivery system:
  1. Successful delivery of the stent in the abdominal aorta and exclusion or treatment of abdominal aortic aneurysm.
  2. follow endoleaks type I, III and IV after 30, 180, and 360 days.
  3. Incidence of major adverse events at 180 and 360 days after implantation or at any time.

CONTACTS AND LOCATIONS:
Overall Officials: Álvaro Razuk, Medicine, Principal Investigator — Irmandade da Santa Casa de Misericórdia de São Paulo
Locations (2):
- Brazil (2):
  - Hospital de Caridade, São Francisco do Sul, Santa Catarina
  - Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo

REFERENCES:
- See also: Site sponsor — http://www.scitechmed.com
- See also: Site about the location that will be done the study. Location where the principal investigator works. — http://www.santacasasp.org.br
- See also: National Information System on Ethics in Research involving Human — http://portal2.saude.gov.br/sisnep